CLINICAL TRIAL: NCT04933227
Title: A Phase II, Single-Arm Study to Explore the Efficacy and Safety of Atezolizumab Plus Tiragolumab and Chemotherapy in 1st Line HER2 Negative Unresectable, Recurrent or Metastatic Gastric Cancer or Adenocarcinoma of Gastroesophageal Junction (GEJ)
Brief Title: A Study to Explore the Efficacy and Safety of Atezolizumab Plus Tiragolumab and Chemotherapy in 1st Line HER2 Negative Unresectable, Recurrent or Metastatic Gastric Cancer or Adenocarcinoma of Gastroesophageal Junction (GEJ)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the study after Stage 1; will not proceed with Stage 2.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42913
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Stomach Neoplasms; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — atezolizumab; Tiragolumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezo + Tira + XELOX (Experimental): Atezolizumab plus tiragolumab in combination with XELOX (oxaliplatin and capecitabine) will be administered during Cycles 1-4 (each cycle is 21 days). During Cycle 5 and beyond atezolizumab and tiragolumab will be administered on Day 1 of each 21-day cycle. Participants will receive study treatment until disease progression, unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered intravenously (IV) on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab 600 mg will be administered IV on Day 1 of each 21-day cycle.
Drug: Oxaliplatin — Oxaliplatin 130 mg/m^2 will be administered IV on Day 1 of each 21-day cycle during Cycles 1-4.
Drug: Capecitabine — Capecitabine 1000 mg/m^2/d will be administered orally (PO) twice daily (bid) on Days 1-14 during Cycles 1-4.

SUMMARY:
This study is designed to evaluate the efficacy and safety of atezolizumab plus tiragolumab in combination with capecitabine plus oxaliplatin (XELOX) for first-line treatment in participants with HER2-negative unresectable advanced, recurrent or metastatic gastric cancer (GC) or gastroesophageal junction adenocarcinoma (GEJ AC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (by enrolling center) gastric cancer or adenocarcinoma of GEJ (Siewert I-III)
* Unresectable locally advanced, unresectable recurrent, or metastatic disease that meets the following criteria: a) No prior systemic treatment for advanced disease, b) For patients receiving prior chemoradiotherapy or chemotherapy in the adjuvant or neoadjuvant setting, with an interval of at least 6 months between the final treatment and the diagnosis of advanced disease
* Measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as determined by investigator assessment
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 and TIGIT expression
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >/=3 months
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to refrain from heterosexual intercourse or use contraception, and agreement to refrain from donating eggs
* For men: agreement to refrain from heterosexual intercourse or use contraceptive methods, and agreement to refrain from donating sperm.

Exclusion Criteria:

* HER2-positive by local review, defined as either immunohistochemistry (IHC) score of 3+ or IHC 2+ with amplification proven by in situ hybridization (ISH) as assessed based on pretreatment tumor tissues
* Use of Chinese herbal medicine or Chinese patent medicines to control cancer within 7 days prior to initiation of study treatment
* Higher risk of bleeding or fistula caused by GEJ Siewert I invading adjacent organs
* Symptomatic, untreated, or actively progressing CNS metastases
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Severe chronic or active infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy within 5 years prior to screening, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death
* Any other disease, medical condition, metabolic dysfunction, alcohol or drug abuse or dependence, physical examination finding, clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Prior treatment with CD137 agonists, T-cell co-stimulating, or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-TIGIT therapeutic antibodies
* Treatment with systemic immunostimulatory agents or any investigational therapy within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment
* Known allergy or hypersensitivity to any component of atezolizumab, tiragolumab, capecitabine or oxaliplatin formulations
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in the Full Analysis Set (FAS) Population | Up to approximately 20 months

SECONDARY OUTCOMES:
Duration of Response (DOR) in Responders of the FAS Population | The time from the first occurrence of a confirmed objective response to the first occurrence of disease progression or death from any cause (whichever occurs first) up to approximately 20 months
Progression-free Survival (PFS) in the FAS Population | The time from initiation of study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first) up to approximately 20 months
Overall Survival (OS) in the FAS Population | The time from initiation of study treatment to death due to any cause up to approximately 20 months
Mean Score in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in the FAS Population | Up to approximately 20 months
Change from Baseline in EORTC QLQ-C30 in the FAS Population | Up to approximately 20 months
Mean Score in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire in Gastric Cancer (EORTC QLQ-STO22) in the FAS Population | Up to approximately 20 months
Change from Baseline in EORTC QLQ-STO22 in the FAS Population | Up to approximately 20 months
ORR in a Subgroup Population With PD-L1 and/or TIGIT Positive Expression | Up to approximately 20 months
Duration of Response (DOR) in Responders of a Subgroup Population With PD-L1 and/or TIGIT Positive Expression | The time from the first occurrence of a confirmed objective response to the first occurrence of disease progression or death from any cause (whichever occurs first) up to approximately 20 months
Progression-free Survival (PFS) in a Subgroup Population With PD-L1 and/or TIGIT Positive Expression | The time from initiation of study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first) up to approximately 20 months
Overall Survival (OS) in a Subgroup Population With PD-L1 and/or TIGIT Positive Expression | The time from initiation of study treatment to death due to any cause up to approximately 20 months
Number of Participants With Adverse Events | Up to approximately 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Changzhou First People's Hospital, Changzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University; Medical Oncology, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Anhui Province Cancer Hospital, Hefei
  - Liaoning cancer Hospital & Institute, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).